CLINICAL TRIAL: NCT03791307
Title: Blood Pressure, Autonomic Heart Rate Modulation, Cardiorespiratory Parameters, Functionality and Quality of Life in Hypertensive Women After 16 Weeks of Training Based on the Pilates Method
Brief Title: Effects of Training Based on the Pilates Method on the Blood Pressure of Hypertensive Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: João Luiz Q. Durigan (Other)
Collaborators: Catholic University of Brasília (Other)
Responsible Party: Sponsor-Investigator, João Luiz Q. Durigan, Physical Therapist, Assistant Professor, University of Brasilia
Organization: University of Brasilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAEE: 99221818.9.0000.0029
Record Dates: First submitted 2018-12-18; First posted 2019-01-02 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Pilates method; Blood pressure; Autonomic heart rate modulation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: One researcher will be blinded to the conduct of evaluations and revaluations. One researcher will be blinded for outcomes statistics analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Pilates group (Experimental): This group will perform only exercises based on the traditional Pilates method
  Interventions: Other: Traditional Pilates group
- Modified Pilates group (Experimental): This group will perform exercises based on the Pilates method alternated with active rest periods on treadmill ergometer
  Interventions: Other: Modified Pilates group
- Control group (No Intervention): This group will not perform any physical exercise during the trial period.

INTERVENTIONS:
Other: Traditional Pilates group — The participants will perform only exercises based on the traditional Pilates method, 2 times a week, for 50 minutes, for 16 weeks.
  Arms: Traditional Pilates group
Other: Modified Pilates group — The participants will perform exercises based on the Pilates method alternated with active rest periods on treadmill ergometer, 2 times a week, for 50 minutes, for 16 weeks.
  Arms: Modified Pilates group

SUMMARY:
The main objective of this study is to evaluate and compare the effect of the Pilates method associated with aerobic exercise and the traditional Pilates method on the blood pressure of hypertensive medicated women. In addition, we aim to analyze and compare the chronic effects of training on cardiac autonomic modulation, on cardiorespiratory fitness, functionality and quality of life.

DETAILED DESCRIPTION:
Subjects will be allocated randomly in three groups: (1) Traditional Pilates group, which will perform only exercises based on the traditional Pilates method, (2) Modified Pilates group, which will perform exercises based on the Pilates method alternated with active rest periods on treadmill ergometer, (3) Control group: will not perform any physical exercise during the trial period. The sessions will be performed two times a week, during 16 weeks. Subjects will be evaluated before and after 16 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive women
* Age 30 to 59
* Sedentary or who do not practice any form of physical exercise regularly for at least 6 months
* Make use of antihypertensive medication
* Who have medical clearance for physical exercise

Exclusion Criteria:

* Complaint of pain that influences or makes the performance of the tests / exercises proposed impossible
* Congenital or acquired anomalies of upper limbs and lower limbs
* Presence of musculoskeletal disease or injury that interfere the performance of exercises
* Changes in pharmacological treatment during the experimental period
* Release for physical activity suspended during intervention
* Absence in more than 25% of the exercise sessions

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure | Change from Baseline systolic and diastolic Blood Pressure at 16 weeks
  Systolic and diastolic blood pressure will be measured by 24-hour Ambulatorial Monitoring Blood Pressure, before and after trial period.

SECONDARY OUTCOMES:
Clinical blood pressure | Change from Baseline systolic and diastolic Blood Pressure at 16 weeks
  Clinical assessment of systolic and diastolic blood pressure will be measured by an automatic arm blood pressure monitor after 10 minutes of rest, before and after trial period.
Clinical heart rate | Change from Baseline clinical heart rate at 16 weeks
  Clinical assessment of heart rate will be measured by a heart rate monitor after 10 minutes of rest, before and after trial period.
Autonomic heart rate modulation | Change from Baseline autonomic heart rate modulation at 16 weeks
  Autonomic heart rate modulation will be assessed by the heart rate variability method using a heart rate monitor, before and after trial period.
Ventilatory threshold measured by the cardiopulmonary exercise test | Change from baseline and at 16 weeks
  The ventilatory threshold will be measured by the cardiopulmonary exercise test. An ergospirometric exercise test will be performed, consisting of increasing loads, with no pauses between the stages until exhaustion of the volunteer. The examination will be performed in a treadmill with ergospirometric and electrocardiographic analysis.
Analysis of the quality of life | Change from Baseline quality of life at 16 weeks
  Quality of life will be analyzed by means of the questionnaire World Health Organization Quality Of Life/Bref (WHOQOL/bref). The questionnaire has twenty-six questions that involve different aspects of daily life and deal with four domains of quality of life: physical, psychological, environmental and social relations. The response is represented by scores ranging from one to five, with the worst score being one and the best score being five. The results of the domains have values between zero and one hundred, with the worst being the closest to zero and the best the closest to one hundred, thus, a value equal to 50 for a given domain can be considered median for that domain.
Flexibility | Change from Baseline flexibility at 16 weeks
  Flexibility will be analyzed by bank of wells test, before and after trial period.
Strength | Change from Baseline strength at 16 weeks
  Strength will be analyzed by hydraulic handgrip dynamometer, before and after trial period.
Speed to lift from a sitting position | Change from Baseline speed at16 weeks
  Speed to lift from a sitting position will be evaluated by a stopwatch, before and after trial period.
Speed to lift from a layered position | Change from Baseline speed at 16 weeks
  Speed to lift from a layered position will be evaluated by a stopwatch, before and after trial period
Speed to put on and tie his shoes | Change from Baseline speed at 16 weeks
  Speed to put on and tie his shoes will be evaluated by a stopwatch, before and after trial period.
Body weight | Change from Baseline body weight at 16 weeks
  Body weight will be measured using a digital scale, before and after trial period.
Height | Change from Baseline at 16 weeks
  Height will be measured using a stadiometer.
Body Mass Index | Change from Baseline body mass index at 16 weeks
  Will be analyzed as weight divided by height squared.
Circumference measurements | Change from Baseline circumference measurements at 16 weeks
  Will be analyzed the circumference of hip, waist, neck, abdomen, before and after trial period.

CONTACTS AND LOCATIONS:
Overall Officials: João LQ Durigan, PhD, Study Director — University of Brasilia
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martins-Meneses DT, Antunes HK, de Oliveira NR, Medeiros A. Mat Pilates training reduced clinical and ambulatory blood pressure in hypertensive women using antihypertensive medications. Int J Cardiol. 2015 Jan 20;179:262-8. doi: 10.1016/j.ijcard.2014.11.064. Epub 2014 Nov 6. PMID 25464462
- [Background] Carpio-Rivera E, Moncada-Jimenez J, Salazar-Rojas W, Solera-Herrera A. Acute Effects of Exercise on Blood Pressure: A Meta-Analytic Investigation. Arq Bras Cardiol. 2016 May;106(5):422-33. doi: 10.5935/abc.20160064. Epub 2016 May 6. PMID 27168471
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Background] Gonzales AI, Nery T, Fragnani SG, Pereira F, Lemos RR, Bezerra PP, Haas P. Pilates Exercise for Hypertensive Patients: A Review of the Literature. Altern Ther Health Med. 2016 Sep;22(5):38-43. PMID 27622959
- [Background] Malachias MV. 7th Brazilian Guideline of Arterial Hypertension: Presentation. Arq Bras Cardiol. 2016 Sep;107(3 Suppl 3):0. doi: 10.5935/abc.20160140. No abstract available. PMID 27819379
- [Background] Niskanen JP, Tarvainen MP, Ranta-Aho PO, Karjalainen PA. Software for advanced HRV analysis. Comput Methods Programs Biomed. 2004 Oct;76(1):73-81. doi: 10.1016/j.cmpb.2004.03.004. PMID 15313543
- [Background] Pescatello LS, MacDonald HV, Lamberti L, Johnson BT. Exercise for Hypertension: A Prescription Update Integrating Existing Recommendations with Emerging Research. Curr Hypertens Rep. 2015 Nov;17(11):87. doi: 10.1007/s11906-015-0600-y. PMID 26423529
- [Background] Prinsloo GE, Rauch HG, Derman WE. A brief review and clinical application of heart rate variability biofeedback in sports, exercise, and rehabilitation medicine. Phys Sportsmed. 2014 May;42(2):88-99. doi: 10.3810/psm.2014.05.2061. PMID 24875976
- [Background] Rtveladze K, Marsh T, Webber L, Kilpi F, Levy D, Conde W, McPherson K, Brown M. Health and economic burden of obesity in Brazil. PLoS One. 2013 Jul 11;8(7):e68785. doi: 10.1371/journal.pone.0068785. Print 2013. PMID 23874763
- [Background] Thompson PD, Buchner D, Pina IL, Balady GJ, Williams MA, Marcus BH, Berra K, Blair SN, Costa F, Franklin B, Fletcher GF, Gordon NF, Pate RR, Rodriguez BL, Yancey AK, Wenger NK; American Heart Association Council on Clinical Cardiology Subcommittee on Exercise, Rehabilitation, and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism Subcommittee on Physical Activity. Exercise and physical activity in the prevention and treatment of atherosclerotic cardiovascular disease: a statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity). Circulation. 2003 Jun 24;107(24):3109-16. doi: 10.1161/01.CIR.0000075572.40158.77. No abstract available. PMID 12821592
- [Background] Weber MA, Schiffrin EL, White WB, Mann S, Lindholm LH, Kenerson JG, Flack JM, Carter BL, Materson BJ, Ram CV, Cohen DL, Cadet JC, Jean-Charles RR, Taler S, Kountz D, Townsend RR, Chalmers J, Ramirez AJ, Bakris GL, Wang J, Schutte AE, Bisognano JD, Touyz RM, Sica D, Harrap SB. Clinical practice guidelines for the management of hypertension in the community: a statement by the American Society of Hypertension and the International Society of Hypertension. J Clin Hypertens (Greenwich). 2014 Jan;16(1):14-26. doi: 10.1111/jch.12237. Epub 2013 Dec 17. No abstract available. PMID 24341872
- [Background] Xhyheri B, Manfrini O, Mazzolini M, Pizzi C, Bugiardini R. Heart rate variability today. Prog Cardiovasc Dis. 2012 Nov-Dec;55(3):321-31. doi: 10.1016/j.pcad.2012.09.001. PMID 23217437
- [Derived] da Silva Almeida I, de Souza Andrade L, de Sousa AMM, Junior GC, Turri-Silva N, Cunha Nascimento DD, Mota YL, Durigan JLQ. The Effect of Mat Pilates Training Combined With Aerobic Exercise Versus Mat Pilates Training Alone on Blood Pressure in Women With Hypertension: A Randomized Controlled Trial. Phys Ther. 2022 Feb 1;102(2):pzab258. doi: 10.1093/ptj/pzab258. PMID 35084038